CLINICAL TRIAL: NCT02699398
Title: Domiciliary VR Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Pompeu Fabra (Other)
Collaborators: Hospital del Mar (Other); Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Paul Verschure, PhD, Universitat Pompeu Fabra
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAL-2008-1-1191
Record Dates: First submitted 2016-02-25; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Hemiparesis; Functional Independence; Movement Disorder; Stroke
MeSH Terms: conditions — Paresis; Movement Disorders; Stroke

ARMS (2):
- VR-based therapy (Experimental): 3 weeks of home-based treatment for motor training using a virtual reality rehabilitation setup.
  Interventions: Behavioral: Domiciliary VR-based motor rehabilitation
- Control (Active Comparator): 3 weeks of home-based occupational therapy for motor training.
  Interventions: Behavioral: Domiciliary occupational therapy for motor rehabilitation

INTERVENTIONS:
Behavioral: Domiciliary VR-based motor rehabilitation — 3 weeks, 1 to 3 sessions a day, 20min per sessions, of physical therapy using a VR gaming system.
  Arms: VR-based therapy
Behavioral: Domiciliary occupational therapy for motor rehabilitation — 3 weeks, 1 to 3 sessions a day, 20min per sessions, of physical therapy using a VR gaming system.
  Arms: Control

SUMMARY:
The purpose of this study is to determine whether domiciliary VR-based telerehabilitation is superior than domiciliary occupational therapy for inducing functional gains, enhancing corticospinal excitability, and cortical reorganization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Hemorrhagic or ischemic stroke
* Subject had the stroke more than 12 months ago.
* Subject presents mild-to-moderate upper-limbs hemiparesis (Proximal Medial Research Council Scale>2) secondary to a first-ever stroke.
* Age between 45 and 85 years old.
* Subject has previous experience using the RGS system in the clinic.

Exclusion Criteria:

* Subject presents a major cognitive impairment (Mini-Mental State Evaluation> 22).

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2011-11; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Change in motor function for activities of daily living as measured by Chedoke Arm Hand Inventory clinical | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.

SECONDARY OUTCOMES:
Change in depression as measured by the Hamilton scale | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in motor function as measured by the Medical Research Council scale | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in spasticity for the upper arms as measured by the Ashworth scale | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in cognitive function as measured by the Mini-mental State Evaluation test | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in Grip Force as measured by a grip dynamometer | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in shoulder pain as measured by the Visual Analog Assessment scale | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.
Change in motor function as measured by the upper extremity Fugl-Meyer Assessment | At baseline, at 3-weeks (after intervention), and at 12-weeks follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Verschure, PhD, Principal Investigator — Synthetic Perceptive, Emotive and Cognitive Systems group, Department of Information and Communication Technologies at the Universitat Pompeu Fabra (UPF).

REFERENCES:
- [Derived] Ballester BR, Nirme J, Camacho I, Duarte E, Rodriguez S, Cuxart A, Duff A, Verschure PFMJ. Domiciliary VR-Based Therapy for Functional Recovery and Cortical Reorganization: Randomized Controlled Trial in Participants at the Chronic Stage Post Stroke. JMIR Serious Games. 2017 Aug 7;5(3):e15. doi: 10.2196/games.6773. PMID 28784593